CLINICAL TRIAL: NCT01972542
Title: The Usefulness of Postprandial Triglyceride for Assessment of Cardiovascular Risk in Healthy People, Impaired Glucose Tolerance and Type 2 Diabetes
Brief Title: The Usefulness of Postprandial Triglyceride for Assessment of Cardiovascular Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Soo Lim, Professor, Seoul National University Bundang Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: SNUBH-ENDO4
Record Dates: First submitted 2013-10-23; First posted 2013-10-30 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-10

CONDITIONS: Diabetes; Prediabetes
Keywords: Postprandial period; triglyceride; Diabetes mellitus, type 2; Prediabetic state
MeSH Terms: conditions — Diabetes Mellitus; Prediabetic State; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Type 2 DM (Active Comparator): Intervention : Oral fat tolerance test
  well or moderately controlled type 2 diabetes mellitus (HbA1c < 10%) No dipeptidyl peptidase-4 -inhibitor, Glucagon-like peptide-1 agonist, thiazolidinediones
  Interventions: Dietary Supplement: Oral fat tolerance test
- Prediabetes (Active Comparator): Intervention : Oral fat tolerance test
  Glucose 140-199 mg/dL after 75g oral glucose tolerance test HbA1c 5.7-6.4%
  Interventions: Dietary Supplement: Oral fat tolerance test
- Normal glucose tolerance (Sham Comparator): Intervention : Oral fat tolerance test
  No impaired fasting glucose and impaired glucose tolerance
  Interventions: Dietary Supplement: Oral fat tolerance test

INTERVENTIONS:
Dietary Supplement: Oral fat tolerance test

SUMMARY:
The hypertriglyceridemia at fasting status has been known to be an important risk factor for cardiovascular disease (CVD). Recently, postprandial triglyceride (TG) levels draw an attention as a superior predictor of CVD because of non-fasting state for more than 12 hours and importance of triglyceride-rich lipoprotein.

We aim to investigate the relationship of postprandial triglyceride after fat tolerance test and intima-medial thickness and to suggest normal reference of postprandial triglyceride after fat tolerance test. In addition, we evaluate the correlation of postprandial triglyceride and incretin secretion after fat tolerance test Ultimately, we want to estimate clinical importance of postprandial triglyceride in assessment of cardiovascular risk.

ELIGIBILITY:
Inclusion Criteria:

* age : 19 ~ 70 yrs
* Type 2 diabetes : HbA1c <10%
* Prediabetic state : HbA1c 5.7~6.4%

Exclusion Criteria:

* Type 1 diabetes, secondary diabetes
* dipeptidyl peptidase-4 -inhibitor, glucagon-like peptide-1 agonist, thiazolidinediones users
* Thyroid disease with abnormal thyroid function test
* Liver disease with abnormal liver function test
* severe kidney disease
* pregnant or lactating women
* current smoker
* severe obesity

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-06; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Changes of Triglyceride | 8 hours
  Blood sample : drawn by a catheter before the meal and every 1 hour after meal over the 8-hour period

SECONDARY OUTCOMES:
Changes of incretin | 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Soo Lim, MD, MPH, PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, South Korea